CLINICAL TRIAL: NCT07170917
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Phase 2 Study of Brivekimig Followed by a Maintenance Period in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Brivekimig for the Treatment of Moderate to Severe Hidradenitis Suppurativa
Acronym: BRIGHTEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI19220; 2025-522333-61-00 (Registry Identifier: CTIS); U1111-1318-3453 (Other: WHO ICTRP)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Brivekimig dose regimen A (Experimental): Participants will receive Brivekimig dose regimen A.
  Interventions: Drug: Brivekimig
- Brivekimig dose regimen B (Experimental): Participants will receive Brivekimig dose regimen B.
  Interventions: Drug: Brivekimig
- Brivekimig dose regimen C (Experimental): Participants will receive Brivekimig dose regimen C.
  Interventions: Drug: Brivekimig
- Placebo (Placebo Comparator): Participants will receive Brivekimig matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brivekimig — * Pharmaceutical form: Solution for injection in vial
  * Route of administration: Subcutaneous injection
  Other Names: SAR442970
  Arms: Brivekimig dose regimen A; Brivekimig dose regimen B; Brivekimig dose regimen C
Drug: Placebo — * Pharmaceutical form: Solution for injection in vial
  * Route of administration: Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a Phase 2b, global, multicenter, sequential, randomized, double-blind, placebo-controlled, parallel group, dose-ranging study in participants with moderate to severe hidradenitis suppurativa.

The purpose of this study is to assess the efficacy and safety of brivekimig in a dose-ranging study of participants with moderate to severe HS.

Study details include:

The study duration (per participant) will be up to approximately 60 weeks for participants not transitioning into the long-term extension (LTE) study and will be up to approximately 52 weeks for participants transitioning into the LTE study.

The randomized treatment duration will be up to approximately 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate to severe hidradenitis suppurativa (HS) for at least 6 months prior to Baseline
* Participants must have HS lesions present in at least 2 distinct anatomic areas (eg, left and right axilla; or left axilla and left inguinocrural fold), one of which must be Hurley Stage II or Hurley Stage III.
* Participant must have had an inadequate response to a trial of an oral antibiotic for treatment of HS, exhibited recurrence after discontinuation of antibiotics, demonstrated intolerance to antibiotics, or has a contraindication to oral antibiotics for treatment of their HS as assessed by the Investigator through participant interview and review of medical history.
* Participants must be either biologic-naive or biologic-experienced.
* Participant must have a total abscess and inflammatory nodule (AN) count of ≥5 at the Baseline visit.
* Participant must have a draining tunnel count of ≤20 at the Baseline visit.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any other active skin disease or condition (eg, bacterial, fungal, or viral infection) that may interfere with assessment of HS
* History of recurrent or recent serious infection
* Known history of significant immunosuppression
* History of solid organ transplant or stem cell transplant
* History of splenectomy
* History of moderate to severe congestive heart failure.
* History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease
* Participants with a history of malignancy or lymphoproliferative disease other than adequately treated or nonmetastatic squamous cell carcinoma of the skin that was excised and completely cured or nonmetastatic basal cell carcinoma of the skin that was excised and completely cured
* History of any other condition which, in the opinion of the Investigator, would put the participant at risk by participation in the protocol
* Active suicidality and therefore significant suicide risk, as judged by the Investigator
* A history of an Adverse Event (AE) attributed to or related to anti-TNF therapy (examples include, but are not limited, to serum sickness or anaphylaxis) for an HS or non-HS indication that would contraindicate readministration of an anti-TNF class therapy
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* History (within last 2 years prior to Baseline visit) of prescription drug or substance abuse, including alcohol, considered significant by the Investigator

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-04-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) is defined as ≥75% reduction from Baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) is defined as ≥50% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining tunnel count.
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 90 (HiSCR90) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 90 (HiSCR90) is defined as ≥90% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining tunnel count.
Change from Baseline in draining tunnel count at Week 16. | From Baseline to Week 16
Change in absolute score from Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) at Week 16 | From Baseline to Week 16
  The determination of IHS4 requires counting the inflammatory nodules, abscesses and draining tunnels and multiplying each by a specific coefficient. A high score signifies severe disease.
Percentage of participants achieving response on the Hidradenitis Suppurativa Skin Pain Numeric Rating Scale from the HS Symptom Assessment Questionnaire (HS-SAQ skin pain NRS) at week 8 | From Baseline to Week 8
  The Hidradenitis Suppurativa Symptom Assessment Questionnaire (HS-SAQ) is a 7-item scale comprising unidimensional numeric rating scale (NRS) items assessing symptoms of HS. The HS-SAQ Skin Pain is based on worst skin pain in a 24-hour recall period (daily assessment is averaged over 7-day period). HS-SAQ skin pain NRS response is defined as ≥3-unit reduction from baseline in the weekly average of daily HS-SAQ Skin Pain NRS.
Change from Baseline in Hidradenitis Suppurativa Quality of Life (HiSQOL) total score at Week 16. | From Baseline to Week 16
  The Hidradenitis Suppurativa Quality of Life is a 17-item content-validated questionnaire with a 7-day recall period. It is scored by summing items to create a total score (0 to 68) with higher score indicating more severe impact on QoL.
Change from Baseline in Dermatology Life Quality Index (DLQI) total score at Week 16. | From Baseline to Week 16
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology specific health related quality of life (HRQoL) instrument. Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Number of participants with treatment-emergent adverse events (TEAE), serious adverse events (SAE) and laboratory anomalies. | Up to End of Study (approximately 60 weeks)
Serum brivekimig concentration throughout the study. | Up to End of Study (approximately 60 weeks)
Incidence of treatment-emergent (TE) anti-drug antibody responses. | Up to End of Study (approximately 60 weeks)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (9):
  - Northridge Clinical Trials - Northridge- Site Number : 8400005, Northridge, California
  - FXM Clinical Research - Miami- Site Number : 8400017, Miami, Florida
  - FXM Clinical Research Miramar, LLC - Site Number: 8400004, Miramar, Florida
  - Advanced Medical Research - Atlanta- Site Number : 8400011, Atlanta, Georgia
  - Georgia Skin & Cancer Clinic- Site Number : 8400009, Savannah, Georgia
  - Louisiana Dermatology Associates- Site Number : 8400006, Baton Rouge, Louisiana
  - Clinical Partners- Site Number : 8400002, Johnston, Rhode Island
  - Alliance for Multispecialty Research - Myrtle Beach- Site Number : 8400018, Myrtle Beach, South Carolina
  - Alpine Research Association- Site Number : 8400008, Layton, Utah
- Alfred Hospital - Site Number: 0360002, Melbourne, Victoria, Australia
- Canada (3):
  - Interior Dermatology Centre - Site Number: 1240003, Kelowna, British Columbia
  - Lima's Excellence in Allergy and Dermatology Research (LEADER) Inc., Hamilton, Ontario
  - Investigational Site Number : 1240009, Toronto, Ontario
- Chile (4):
  - Investigational Site Number: 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number: 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number: 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number: 1520005, Santiago, Reg Metropolitana de Santiago
- China (2):
  - Investigational Site Number : 1560002, Chengdu
  - Investigational Site Number : 1560001, Guangzhou
- Czechia (4):
  - Investigational Site Number: 2030002, Ostrava
  - Investigational Site Number: 2030003, Ostrava
  - Investigational Site Number: 2030001, Prague
  - Investigational Site Number: 2030004, Prague
- Investigational Site Number : 2760008, Bramsche, Germany
- Investigational Site Number : 3480004, Székesfehérvár, Hungary
- Israel (2):
  - Investigational Site Number: 3760002, Jerusalem
  - Investigational Site Number: 3760001, Tel Aviv
- Japan (3):
  - Meiwa Hospital, Nishinomiya, Hyōgo
  - University of the Ryukyus Hospital - Site Number: 3920002, Nishihara, Okinawa
  - Nihon University Itabashi Hospital, Tokyo
- Investigational Site Number: 6160003, Lodz, Lódzkie, Poland
- Spain (4):
  - Investigational Site Number: 7240003, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number: 7240002, Manises, Valencia
  - Investigational Site Number : 7240007, Granada
  - Investigational Site Number: 7240001, Madrid
- United Kingdom (2):
  - Investigational Site Number : 8260008, London, England
  - Investigational Site Number : 8260006, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI19220 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26950&tenant=MT_SNY_9011